CLINICAL TRIAL: NCT03265483
Title: Effect of Magnesium Treatment on Vitamin D Resistance
Brief Title: Magnesium Treatment on Vitamin D Metabolism in Participants Completed Personalized Prevention of Colorectal Cancer Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Martha Shrubsole, Research rofessor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 100106b
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
Keywords: Personalized prevention trial; Magnesium; Vitamin D metabolism and synthesis; Magnesium-vitamin D interaction
MeSH Terms: conditions — Colorectal Neoplasms | interventions — magnesium diglycinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium treatment (Active Comparator): Participants will be assigned to magnesium glycinate
  Interventions: Dietary Supplement: Magnesium glycinate
- Placebo (Placebo Comparator): Participants will be assigned to placebo group
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium glycinate — Oral administration of magnesium glycinate daily for 12 weeks
  Arms: Magnesium treatment
Dietary Supplement: Placebo — Oral administration of identical-appearing placebo daily for 12 weeks
  Arms: Placebo

SUMMARY:
One striking observation is that a large portion of the inter-person variation in serum 25-hydroxyvitamin D (25(OH)D) levels is unexplained. In vitro and in vivo studies indicate vitamin D synthesizing and metabolizing enzymes are Mg-dependent. Magnesium (Mg) supplementation substantially reversed the resistance to vitamin D treatment in patients with magnesium-dependent vitamin-D-resistant rickets. The investigators reported in 2013 from observational studies conducted in the general US population that Mg intake significantly interacted with vitamin D intake in affecting vitamin D status as well as interacted with serum 25(OH)D in risk of cardiovascular disease mortality and, maybe, colorectal cancer mortality. The potential interaction between Mg and vitamin D was supported by two subsequent studies, including a Finnish cohort study and a mouse study.

In the parent study (Personalized Prevention of Colorectal Cancer Trial, NCT01105169), the investigators proposed to measure blood concentration of total 25(OH)D as a secondary aim using Elisa approach. However, following the novel finding of Mg-vitamin D interaction published by the investigators in 2013, they submitted a separate grant application to NCI which was funded in 2014. In the new study, the investigators proposed to use a LC-MS approach, which is more accurate and specific than an Elisa method, to measure 5 vitamin D metabolites. This new ancillary study allows the investigators to evaluate whether Mg supplementation differentially affects vitamin D synthesis and metabolism dependent on baseline serum 25(OH)D levels using existing biospecimens collected in our double-blind placebo-controlled randomized chemoprevention trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participants from our parent study (Personalized Prevention of Colorectal Cancer Trial, NCT#01105169, IRB#100106);
2. Participants who had completed the above study before the time of the sample selection (October 2015);
3. Participants consent to store/share samples for future research in colorectal tumors.

Exclusion Criteria:

1. Participants cannot provide their blood samples in the parent study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Sun E, Zhu X, Ness RM, Murff HJ, Sun S, Yu C, Fan L, Azcarate-Peril MA, Shrubsole MJ, Dai Q. Magnesium treatment increases gut microbiome synthesizing vitamin D and inhibiting colorectal cancer: results from a double-blind precision-based randomized placebo-controlled trial. Am J Clin Nutr. 2025 Nov;122(5):1185-1194. doi: 10.1016/j.ajcnut.2025.09.011. Epub 2025 Sep 12. PMID 40946805
- [Derived] Zhu X, Borenstein AR, Zheng Y, Zhang W, Seidner DL, Ness R, Murff HJ, Li B, Shrubsole MJ, Yu C, Hou L, Dai Q. Ca:Mg Ratio, APOE Cytosine Modifications, and Cognitive Function: Results from a Randomized Trial. J Alzheimers Dis. 2020;75(1):85-98. doi: 10.3233/JAD-191223. PMID 32280092
- [Derived] Dai Q, Zhu X, Manson JE, Song Y, Li X, Franke AA, Costello RB, Rosanoff A, Nian H, Fan L, Murff H, Ness RM, Seidner DL, Yu C, Shrubsole MJ. Magnesium status and supplementation influence vitamin D status and metabolism: results from a randomized trial. Am J Clin Nutr. 2018 Dec 1;108(6):1249-1258. doi: 10.1093/ajcn/nqy274. PMID 30541089

RESULTS

PARTICIPANT FLOW:
Groups:
- Magnesium Glycinate Supplements: Participants will be assigned to magnesium glycinate
  Magnesium glycinate: Oral administration of magnesium glycinate daily for 12 weeks
Period: Overall Study
Arm/Group | Magnesium Glycinate Supplements | Placebo
Started | 87 | 93
Completed | 87 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is an NCI-funded ancillary study nested in the parent study (registered at clinicaltrials.gov as NCT01105169). For the current study, 180 participants who had completed the parent study by October 2015 were selected, including 87 participants in the treatment arm and 93 in the placebo arm. Based on the proposal, we compared the vitamin D metabolites between the two arms (magnesium treatment vs placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Glycinate Supplements | Placebo | Total
Number analyzed (Participants) | 87 | 93 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.3) | 61.7 (8.3) | 61.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 48 | 90
  Male | 45 | 45 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 85 | 92 | 177
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Comparisons of the Changes of Blood 25-Hydroxyvitamin D3 (25(OH)D3) Between Magnesium Treatment and Placebo Arm, Stratified by the Baseline 25-hydroxyvitamin D (25(OH)D) Levels
Description: 25(OH)D3 was extracted from plasma by liquid extraction and measured by using a novel liquid chromatography-mass spectrometry (LC-MS) method.
  The baseline 25(OH)D were measured by: the baseline value of 25(OH)D2 + the baseline value of 25(OH)D3.
  The changes of 25(OH)D3 were measured as: the post-treatment value of 25(OH)D3 (at Week 12) - the pre-treatment value of 25(OH)D3 (at baseline).
Time Frame: 12 weeks
Population: What we include in Rows are not estimates in subgroups, but model-based predictions given specific values of baseline 25-hydroxyvitamin D (25(OH)D) levels. The mean prediction and its standard error are calculated using model coefficient estimates and its variance-covariance matrix, and the sample size is equal to the number of subjects used to fit the model, i.e., overall number of participants analyzed.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- The Changes in Magnesium Treatment Arm: Participants in magnesium supplements: the changes of 25(OH)D3 were measured as: the post-treatment value of 25(OH)D3 (at Week 12) - the pre-treatment value of 25(OH)D3 (at baseline).
- The Changes in Placebo Arm: Participants in placebo: the changes of 25(OH)D3 were measured as: the post-treatment value of 25(OH)D3 (at Week 12) - the pre-treatment value of 25(OH)D3 (at baseline).
Arm/Group | The Changes in Magnesium Treatment Arm | The Changes in Placebo Arm
Number analyzed (Participants) | 87 | 93
ng/mL
  Baseline 25(OH)D=30 | 32.20 (1.56) | 29.41 (1.61)
  Baseline 25(OH)D=20 | 30.95 (2.18) | 29.37 (2.08)
  Baseline 25(OH)D=40 | 29.76 (1.84) | 30.31 (1.80)
  Baseline 25(OH)D=50 | 24.89 (2.74) | 31.76 (2.00)

2. Primary Outcome: Comparisons of the Changes of Blood 25-Hydroxyvitamin D2 (25(OH)D2) Between Magnesium Treatment and Placebo Arm, Stratified by the Baseline 25-hydroxyvitamin D (25(OH)D) Levels
Description: 25(OH)D2 was extracted from plasma by liquid extraction and measured by using a novel liquid chromatography-mass spectrometry (LC-MS) method.
  The baseline 25(OH)D were measured by: the baseline value of 25(OH)D2 + the baseline value of 25(OH)D3.
  The changes of 25(OH)D2 were measured as: the post-treatment value of 25(OH)D2 (at Week 12) - the pre-treatment value of 25(OH)D2 (at baseline).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL (log-transformed)
Groups:
- The Changes in Magnesium Treatment Arm: Participants in magnesium supplements: the changes of 25(OH)D2 were measured as: the post-treatment value of 25(OH)D2 (at Week 12) - the pre-treatment value of 25(OH)D2 (at baseline).
- The Changes in Placebo Arm: Participants in placebo: the changes of 25(OH)D2 were measured as: the post-treatment value of 25(OH)D2 (at Week 12) - the pre-treatment value of 25(OH)D2 (at baseline).
Arm/Group | The Changes in Magnesium Treatment Arm | The Changes in Placebo Arm
Number analyzed (Participants) | 87 | 93
ng/mL (log-transformed)
  Baseline 25(OH)D=20 | -2.22 (0.57) | -1.65 (0.55)
  Baseline 25(OH)D=30 | -1.94 (0.45) | -1.38 (0.46)
  Baseline 25(OH)D=40 | -1.68 (0.44) | -2.13 (0.45)
  Baseline 25(OH)D=50 | -1.43 (0.55) | -3.56 (0.57)

3. Primary Outcome: Comparisons of the Changes of Blood 24,25-dihydroxyvitamin D3 (24,25(OH)2D3) Between Magnesium Treatment and Placebo Arm, Stratified by the Baseline 25-hydroxyvitamin D (25(OH)D) Levels
Description: 24,25(OH)2D3 was extracted from plasma by liquid extraction and detected by using a novel liquid chromatography-mass spectrometry (LC-MS) method.
  The baseline 25(OH)D were measured by: the baseline value of 25(OH)D2 + the baseline value of 25(OH)D3.
  The changes of 24,25(OH)2D3 were measured as: the post-treatment value of 24,25(OH)2D3 (at Week 12) - the pre-treatment value of 24,25(OH)2D3 (at baseline).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- The Changes in Magnesium Treatment Arm: Participants in magnesium supplements: the changes of 24,25(OH)2D3 were measured as: the post-treatment value of 24,25(OH)2D3 (at Week 12) - the pre-treatment value of 24,25(OH)2D3 (at baseline).
- The Changes in Placebo Arm: Participants in placebo: the changes of 24,25(OH)2D3 were measured as: the post-treatment value of 24,25(OH)2D3 (at Week 12) - the pre-treatment value of 24,25(OH)2D3 (at baseline).
Arm/Group | The Changes in Magnesium Treatment Arm | The Changes in Placebo Arm
Number analyzed (Participants) | 87 | 93
ng/mL
  Baseline 25(OH)D=20 | 4.35 (0.41) | 3.96 (0.39)
  Baseline 25(OH)D=30 | 4.31 (0.32) | 3.90 (0.32)
  Baseline 25(OH)D=40 | 3.47 (0.32) | 3.91 (0.32)
  Baseline 25(OH)D=50 | 2.12 (0.44) | 3.97 (0.36)

ADVERSE EVENTS:
Groups:
- Magnesium Supplements: Participants in magnesium treatment: oral administration of magnesium glycinate daily for 12 weeks
- Placebo: Participants in placebo: oral administration of identical-appearing placebo daily for 12 weeks
Arm/Group | Magnesium Supplements | Placebo
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/93
Other Adverse Events (participants affected / at risk) | 0/87 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No